CLINICAL TRIAL: NCT06367725
Title: Pharmacokinetics of Dexamethasone in Childhood ALL and Reduction in Bone Mineral Density
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 1-10-72-122-23
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about, the systemic exposure to dexamethason in childhood acute lymphatic leukemia (ALL). The main questions it aims to answer are:

* How does the intake of dexamethasone correlate with systemic exposure to dexamethason?
* Does systemic exposure to dexamethasone correlate with a reduction in bone mineral density?

Participants will:

* Continue to receive the best available therapy for ALL in Western Europe.
* Have blood samples taken from their central line to measure dexamethasone levels.
* When standard lumbar punctures are done as part of treatment, a sample of cerebrospinal fluid will also be taken to analyze dexamethasone.
* Visit the clinic four times for a DXA scans to measure bone density and vertebral fracture assessment: within three weeks of starting treatment, six months after starting treatment, one month after finishing treatment, and one year after finishing treatment. Biomarkers related to bone health will also be collected on these days. Additionally, participants will fill out questionnaires to track their daily physical activity levels.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of acute lymphoblastic leukaemia
* Age 1-17.9 years

Exclusion Criteria:

* Down syndrome

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and adolescents diagnosed with ALL and treated according to the established and approved treatment protocol in Denmark
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration Curve (AUC) of Dexamethasone | Repeated during induction, with AUC measurements on days 3, 4, and 15. Blood samples taken before dosing, and after 1, 2, 4, and 6 hours
  Blood samples

SECONDARY OUTCOMES:
Mineral bone density by DXA-scan | Within 3 weeks of treatment initiation, 6 months after treatment initiation, one month after ended treatment and 1 year after end of treatment.
  DXA-scan
Vertebral fracture assessment (VFA) by DXA-scan | Within 3 weeks of treatment initiation, 6 months after treatment initiation, one month after ended treatment and 1 year after end of treatment.
  DXA-scan
Dexamethasone in cerebrospinal fluid | When lumbar punctures are performed according to standard treatment during induction
  Comparing measurements of dexamethasone in blood and cerebrospinal fluid

OTHER OUTCOMES:
Physical activity questionnaire | Within 3 weeks of treatment initiation, 6 months after treatment initiation, one month after ended treatment and 1 year after end of treatment.
Biomarkers of bone metabolism | Within 3 weeks of treatment initiation, 6 months after treatment initiation, one month after ended treatment and 1 year after end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte K Albertsen, Professor, Principal Investigator — Department of Paediatrics and Adolescent Medicine, Aarhus University Hospital
Locations (4):
- Denmark (4):
  - Department of Paediatrics and Adolescent Medicine, Copenhagen University Hospital Rigshospitalet, Copenhagen, København Ø
  - Department of Paediatrics and Adolescent Medicine, Odense University Hospital, Odense, Odense C
  - Department of Paediatrics and Adolescent Medicine, Aalborg University Hospital, Aalborg
  - Department of Paediatrics and Adolescent Medicine, Aarhus University Hospital, Aarhus N

IPD SHARING:
Plan to Share IPD: No